CLINICAL TRIAL: NCT05664815
Title: Benefit of Cryopreserved Human Amniotic Membrane (hAM) on Oral Mucosal Healing Among Patients With Stage II Maxillomandibular Osteonecrosis Induced by Antiresorptive and/or Anti-angiogenic Therapies: a Phase II Randomized Trial
Brief Title: Human Amniotic Membrane (hAM) for Stage II Maxillomandibular Osteonecrosis Management
Acronym: amniOST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/584
Record Dates: First submitted 2022-10-24; First posted 2022-12-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteonecrosis Due to Drugs, Jaw
MeSH Terms: interventions — cancer procoagulant; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Randomization 3:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of human amniotic membrane (hAM) (Experimental): After conventional/standard treatment, hAM will be applied in a single layer against the bone defect before closure.
  Interventions: Biological: Human Amniotic Membrane
- Conventional/standard treatment (Active Comparator): Conventional/standard surgery.
  Interventions: Other: Conventional/Standard treatment

INTERVENTIONS:
Biological: Human Amniotic Membrane — After conventional/standard treatment, hAM will be applied in a single layer against the bone defect with, if possible, a burial of a few millimeters under the mucous edges.
  With the idea of apprehending a possible dose effect, the hAM will be adapted to the size of the bone/mucous defect, mesenchymal side against the bone.
  For closure after hAM grafting : 2 options are possible:
  Edge-to-edge closure if sufficient mucosal laxity, Edge rapprochement by cross points. If necessary: possible incision of the periosteum to give laxity to the mucosa.
  Other Names: hAM; amnion
  Arms: Application of human amniotic membrane (hAM)
Other: Conventional/Standard treatment — Surgical procedure: Endo-oral approach:
  * Trimming of the mucous edges if they are necrotic or inflamed (granulation tissue)
  * For the bone: either simple sequestrectomy (the mobile sequestered bone is grabbed using forceps); either reaming until bleeding is obtained; either resection with the rongeur; either monobloc resection of the entire necrotic fragment with a saw or with a piezzotome (ultrasound); or a combination of different techniques. Rq: the resection of the necrotic bone (according to the practices of the center) will operate until the appearance of an "apparently healthy" bone (bone bleeding, clean appearance of the bone site)
  * Closure of the mucosa with possible incision of the periosteum to provide laxity: Suture points by points separated in one plane with non-absorbable braided thread of the 3.0 "silk thread" type and round needle.
  Arms: Conventional/standard treatment

SUMMARY:
This study aims to demonstrate, during the first standard surgical management of patients with stage II MRONJ, the effect of the implantation of a cryopreserved hAM on the maxillomandibular bone, on the healing of the oral mucosa.

DETAILED DESCRIPTION:
Medication-Related Osteonecrosis of the Jaw (MRONJ) is a complication of taking anti-tumor (anti-angiogenic) and bone anti-resorptive treatments (biphosphonates, Denosumab) which impact bone healing and renewal capacities, which can lead to bone necrosis. It affects 1 to 10% of patients and is classified into 4 stages.

There is no reference document for their management, which requires antibiotics, local antiseptics and tissue debridement sometimes associated with sequestrectomy. The objective of treatment is very often to obtain healing of the oral mucosa to cover the exposed bone. Without treatment, stage II MRONJ can progress to stage III, with orostoma, pathological fractures and extra-fistula.

The human amniotic membrane (hAM) has poor (even no) immunogenicity and exerts an anti-inflammatory, anti-fibrotic, antimicrobial, antiviral and analgesic effect. It is a source of multipotent stem cells and growth factors that promote tissue regeneration.

A pioneering, non-comparative study reports the use of hAM in MRONJ with very encouraging results in terms of re-epithelialization, absence of pain and infection (Ragazzo 2018). Recently, the same team published a retrospective study where 49 patients (stage 1 to 3) were included, including 27 treated with hAM (Ragazzo 2021). They report a significant improvement in quality of life and pain in the treated group.

hAM would provide a new approach in the treatment of stage II MRONJ by acting on: the quality and speed of mucosal healing, pain, even infection and regeneration of the underlying bone.

This study aims to demonstrate, during the first standard surgical management of patients with stage II MRONJ, the effect of the implantation of a cryopreserved hAM on the maxillomandibular bone, on the healing of the oral mucosa three months after the operation.

In second objectives will be evaluated: pain, complications at the site of healing of the mucosa (erythema, abscess, purulent discharge, diffuse infection of soft tissues (cellulitis), orostoma, suborbital abscess, mandibular fracture), oral health -dental/quality of life and new bone formation at subsequent visits.

ELIGIBILITY:
INCLUSION CRITERIA

* Men and women over the age of 18
* Patient treated in the context of a tumor pathology during which he received treatment with bisphosphonates, Denosumab or anti-angiogenics, and/or, very often, switch of treatment or combination. Current treatment or mention of treatment in patient history
* MRONJ stage II certified clinically and radiologically. Also in the maxilla, stage II MRONJ without bucco-sinus communication after excision of the necrotic bone. Similarly, if a tooth with antral roots must be extracted and creates a bucco-sinus communication, if a MRONJ results, it will be stage II
* Patients with stage II MRONJ of childbearing age with current contraception or patients already postmenopausal
* Signature of the informed consent to participate indicating that the subject has understood the purpose and the procedures required by the study, that he agrees to participate in the study as well as to comply with the requirements and restrictions inherent in this study
* Affiliation to a French social security scheme or beneficiary of such a scheme

NON-INCLUSION CRITERIA

* Life expectancy of less than 6 months assessed by oncologists
* Existence of an evolving cervico-facial neoplasia or an evolving oral neoplastic process informed by oncologists
* History of oral and/or cervico-facial radiotherapy
* Allergy to one of these two antibiotics: amoxicillin-clavulanic acid or clindamycin-metronidazole combination
* Patient contraindicated for surgery due to his state of health, with general anesthesia or local anesthesia.
* MRONJ stage I and stage III
* Stage II MRONJ in patients with only osteoporosis
* Patients receiving treatments that may affect bone and/or mucous tissue as well as their metabolism: Patients on long-term corticosteroid therapy or immunosuppressants
* Patients with other diseases that may affect bone and/or mucous tissue as well as their metabolism: Bone diseases (such as brittle bone disease or Osteogenesis imperfecta, primary bone tumors in the maxilla or mandible (osteosarcoma, sarcoma, rhabdomyosarcoma ,…), any other malignant bone tumour; metabolic diseases with bone repercussions (Paget's disease, osteomalacia,…)
* Patients of childbearing age without contraception
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject not affiliated to a social security scheme
* Patient under guardianship, curatorship or imprisonment
* Patient who notified his refusal to participate in the research
* Patient who participates in another clinical research

EXCLUSION CRITERIA

* During surgery: Discovery of an interrupting MRONJ with damage to the basilar edge (which corresponds to stage III).
* During surgery: Following a sequestrectomy discovery of spontaneous or ongoing healing.
* During the inclusion period: Patient to benefit from invasive "dental" surgeries directly related to bone exposure and in conjunction with taking risky molecules (factors favoring the occurrence of MRONJ): dental avulsions, curettage apical granulomas or cysts, endodontic treatments, or alveolar bone procedure (regularization of ridges).
* During the inclusion period: Patient with metastases all over the mandible.
* During the inclusion period: State of health of the patient which deteriorates due to his cancer during the inclusion period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with re-apparition of bone exposure | Between Day 1 post-surgery and Month 3 post-surgery
  Number of patients with re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area

SECONDARY OUTCOMES:
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Day 0 (the day of the surgery) or Day 1 post-surgery
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Visit 1 (7 to 10 days post-surgery)
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Visit 2 (14 to 15 days post-surgery)
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Visit 3 (One month post-surgery),
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Visit 5 (6 months post-surgery)
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
Number of patient with re-opening of the scar / reappearance of the bone exposure added visually during the control visit | Visit 6 (12 months post-surgery)
  Re-apparition of bone exposure visually observed by the surgeon. Clinical examination: reopening of the scar / reappearance of exposed bone / taking a photograph of the treated area
To assess pain with Visual Analogue Scale | Day 0 or Day 1 (if hospitalized patient)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 1 (7 to 10 days post-surgery)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 2 (14 to 15 days post-surgery)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 3 ( 1 Month post-surgery)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 4 (3 Month post-surgery),
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 5 (6 Month post-surgery)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
To assess pain with Visual Analogue Scale | Visit 6 ( 12 Month post-surgery)
  Pain assessed by a Visual Analogue Scale (VAS). This EVA scale will be supplemented by a collection of information on the use of analgesics if necessary. Also patients who would have to take analgesics will fill out a "logbook" which will specify the class of the drug and the dosage.
Proportion of subjects with a complication at the site of mucosal healing | Day 0 or Day 1 post-surgery (if hospitalized patient)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | visit 1 (7 to 10 days post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | Visit 2 (14 to 15 days post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | Visit 3 (Month1 post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | Visit 4 ( 3 Month post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | Visit 5 (6 Month post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
Proportion of subjects with a complication at the site of mucosal healing | Visit 6 (Month 12 post-surgery)
  On examination of the area of interest, during each visit, search for the presence of:
  * Minor complications: pain and/or erythema and/or abscess and/or purulent discharge,
  * Major complications: diffuse soft tissue infection (cellulitis), orostoma, suborbital abscess, mandibular fracture.
quality of life related to oral health | Day 0 or Day +1 post-surgery (if hospitalized patient)
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | Visit1 (7 to10 days post-surgery)
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | Visit 2 (14 to 15 days post-surgery)
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | V3 (Month 1 post-surgery),
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | Visit 4 ( Month 3 post-surgery)
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | Visit 5 (Month 6 post-surgery)
  Oral health impact profile OHIP 14 quality of life score
quality of life related to oral health | Visit 6 (Month 12 post-surgery)
  Oral health impact profile OHIP 14 quality of life score
Proportion of subjects with new bone formation | Visit 4 (Month 3)
  Presence of newly formed bone assessed by cone-beam imaging
Proportion of subjects with new bone formation | Visit 5 (Month 6)
  Presence of newly formed bone assessed by cone-beam imaging

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien LOUVRIER, MD, PhD, Principal Investigator — CHU de Besançon
Locations (5):
- France (5):
  - CHU de Besancon, Besançon
  - CHU Bordeaux Pellegrin, Bordeaux
  - CHU de Dijon, Dijon
  - CHR Metz Thionville, Metz
  - CHU de Reims, Reims